CLINICAL TRIAL: NCT03188302
Title: Evaluation of a New Method for Measuring Stool Consistency, Using a Texture Analyser (TA.XT Express Texture Analyser)
Brief Title: Evaluation of New Method for Measuring Stool Consistency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yakult Honsha European Research Center, ESV (Other)
Collaborators: Harmony Clinical Research BVBA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: YHER16-TAXT
Record Dates: First submitted 2017-06-08; First posted 2017-06-15 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Stool consistency; Texture Analyser; Bristol Stool Form Scale

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Specimen collection (Other): Collection of stool samples
  Interventions: Other: Collection of stool samples

INTERVENTIONS:
Other: Collection of stool samples — The subjects collect stool samples to be used for validation of a new direct measurement of stool consistency. Every stool sample produced during 2 collection periods of approximately 60 hours each have to be collected using the Commode Specimen Collection System (Medline Industries, Inc.). Each collection period starts preferably in the evening (20h00) and ends 3 days later in the morning (08h00). The collected samples must be stored at subject's home in a refrigerator provided by the sponsor until handover to the site staff.

SUMMARY:
This study is designed to validate a new direct method for the measurement of stool consistency, using Texture Analyser. Forty healthy subjects are enrolled in this trial for collection of stool samples. Every stool produced during 2 collection periods of approximately 60 hours each is collected and subjected to the measurement of consistency using Texture Analyser. The stool consistency results are compared with the Bristol Stool Form Scale scores for each stool. The relationships of stool consistency with other stool parameters, bowel habit and sleeping habit are also evaluated.

DETAILED DESCRIPTION:
It is now obvious that the proper functioning of the gastrointestinal tract has a positive effect on the quality of life. Normal bowel habits vary considerably from person to person with regard to frequency of bowel movements, and bulk and consistency of stools. Constipation is the common digestive complaint in European populations, and softening stool consistency can be regarded as beneficial for such population in terms of reducing incidence of hard or lumpy stools .

The Bristol Stool Form Scale (BS) is validated as a surrogate measure for gastrointestinal transit time, and has been also applied to an evaluation of stool consistency. Subjects compare their stool with the BS chart consisting of seven categories and choose one score which has a nearest analog form. The BS has been widely used in the studies to evaluate changes in stool consistency after dietary intervention using probiotics and/or prebiotics. However, there is a lack of evidence in the validity of BS to yield consistent and reproducible estimates of changes in stool consistency over time. In order to obtain a closer estimate of its change, it would be preferred to use a more directly observable and objective parameter or combination of parameters.

From the above mentioned backgrounds, this study is conducted to validate a new direct method for the measurement of stool consistency, using Texture Analyser: TA.XTExpress Texture Analyser (Stable Micro Systems Ltd.).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities.
* Healthy female or male aged 18 years (inclusive) or older.
* Is willing and able to provide at least 3 stool samples during 2 collection periods of approximately 60 hours, to store the samples in appropriate conditions and to return the samples within the required timeframe.
* Is willing and able to complete a diary during the stool collection periods in order to collect information about form of the stools (based on the Bristol Stool Form Scale classification), bowel habit and sleep habit.
* Understands the Dutch or English language (reading, writing, speaking).

Exclusion Criteria:

* Language barrier, mental or legal incapacity, unwillingness or inability to understand or not being able to participate in this trial.
* Is treated (i.e., currently treated, treated within 1 month before inclusion) for constipation, diarrhoea or any other illness, by use of antibiotics or any other treatment with impact on defecation.
* Females of child bearing potential who are pregnant, breast-feeding or intend to become pregnant.
* Is unable to refrain from or anticipates the use of disallowed medications, e.g., antibiotics, laxatives, anti-diarrheal medication.
* Has any history of drug and/or alcohol abuse.
* Any clinically significant disease which in the Investigator's opinion could interfere with the safety of study participants or with the results of the study.
* Participation in another interventional clinical study or receipt of any investigational product within 1 month before visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Stool consistency | Two stool collection periods of approximately 60 hours each
  Stool consistency is measured as force (g) during compression by Texture Analyser. A cylinder probe is put vertically into the object with a constant speed and the force is measured when reaching down to the target (5 mm down from the surface) as an outcome.

SECONDARY OUTCOMES:
Bristol Stool Form Scale score | Two stool collection periods of approximately 60 hours each
  Bristol Stool Form Scale (BS) is for classifying the form of stool into 7 categories scored from 1 to 7; (1) Separate hard lumps like nuts (difficult to pass); (2) Sausage-shaped but lumpy; (3) Like a sausage but with cracks on its surface; (4) Like a sausage or snake, smooth and soft; (5) Soft blobs with clear-cut edges (passed easily); (6) Fluffy pieces with ragged edges, a mushy stool; (7) Watery, no solid pieces, entirely liquid. Subjects choose one of the BS scores which has a nearest analog form with their stools at every defecation.
Stool water content | Two stool collection periods of approximately 60 hours each
  Percentage of water in stool (weight/weight %)
Stool mucin | Two stool collection periods of approximately 60 hours each
  Concentration of mucin in stool
Stool pH | Two stool collection periods of approximately 60 hours each
  Degree of stool pH
Stool metabolites | Two stool collection periods of approximately 60 hours each
  Concentrations of stool metabolites including organic acids
Stool microbiota composition | Two stool collection periods of approximately 60 hours each
  Relative abundance of microbiota species (% of total) in stool
Stool amount | Two stool collection periods of approximately 60 hours each
  Weight (g) of stool produced in each defecation
Bowel habit | Two stool collection periods of approximately 60 hours each
  Presence or absence of straining during evacuation, presence or absence of sensation of remaining stool in the rectum after evacuation
Sleep habit | Two stool collection periods of approximately 60 hours each
  Getting-up time, going-to-bed time and sleeping hours

CONTACTS AND LOCATIONS:
Overall Officials: Ignace Demeyer, Dr., Principal Investigator — Onze-Lieve-Vrouw Hospital Aalst
Locations (1):
- Onze-Lieve-Vrouw Hospital Aalst, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: No